CLINICAL TRIAL: NCT04791904
Title: Predictive Factors for Cranioplasty Complications - A Decade Experience
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Ana Filipa Vaz Ferreira, Principal Investigator, Universidade do Porto
Other Study IDs: 202101
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Decompressive Craniectomy and Cranioplasty
Keywords: Cranioplasty; Surgery Complications; Decompressive Craniectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center, observational retrospective study. This study aims to identify predictive factors of complications for patients submitted to cranioplasty after decompressive craniectomy for all types of etiologies.

All patients submitted to cranioplasty since 2008 will be analyzed.

DETAILED DESCRIPTION:
Patients submitted to cranioplasty since 2008 to 2019 will be retrospectively analyzed.

Will be considered for analysis all cases treated after decompressive craniectomy. Will be excluded patients with incomplete clinical or imaging records.

Main factors determined as a possible influence on complications after cranioplasty will be recorded focusing on patients characteristics, craniectomy characteristics, surgical timing, and cranioplasty materials.

Patients' records will be review by two investigators and data will be verified by a third investigator. records will be anonymously recorded.

ELIGIBILITY:
Inclusion Criteria:

* Cranioplasty surgery
* Previous decompressive craniectomy

Exclusion Criteria:

* Incomplete records (Clinical and Imaging) since craniectomy to 6 months after cranioplasty.
* More than one decompressive craniectomy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients submitted to cranioplasty after decompressive craniectomy between 1 of January of 2008 and 21 of December of 2019.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Surgical Complications | 6 months
  Complications after cranioplasty - symptomatic hemorrhage, infection, re-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Silva, MD, Study Director — University of Porto, Medicine Faculty
Locations (1):
- Centro Hospitalar Universitário de São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No